CLINICAL TRIAL: NCT00652834
Title: Gastrointestinal Mucosal Findings in Patients Receiving Mycophenolic Acid (MPA) as Demonstrated by Small Bowel Capsule Endoscopy (SBCE)
Brief Title: Small Bowel Capsule Endoscopy Findings in Patients Receiving Cellcept®
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of California, Los Angeles (Other)
Collaborators: Novartis (Industry)
Responsible Party: Principal Investigator, Suphamai Bunnapradist, Principal Investigator, University of California, Los Angeles
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 11-001911
Record Dates: First submitted 2008-04-01; First posted 2008-04-04 (Estimated); Results first posted 2016-03-04 (Estimated); Last update posted 2016-03-04 (Estimated); Status verified 2014-12

CONDITIONS: Gastrointestinal Lesions; Signs and Symptoms, Digestive
Keywords: Renal transplant recipients; Gastrointestinal findings in small bowel capsule endoscopy; Mycophenolic acid; Mycophenolate Mofetil; Mycophenolate Sodium
MeSH Terms: conditions — Signs and Symptoms, Digestive | interventions — Endoscopy; Mycophenolic Acid

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- kidney recipients with GI symptoms (Other): This was a four-week study designed to investigate GI mucosal lesions by SBCE in kidney transplant recipients who were using MMF, and to examine the changes in clinical symptoms and intestinal mucosa lesions 30 days after switching over from MMF to EC-MPS. The patient was switched from MMF to EC-MPS (Myfortic) on the equimola basis.
  Interventions: Procedure: Small bowel capsule endoscopy (SBCE); Drug: myfortic

INTERVENTIONS:
Procedure: Small bowel capsule endoscopy (SBCE) — SBCE will be performed at Day 2 and Day 30.
  Other Names: PillCamEso
Drug: myfortic — switching from mycophenolate mofetil to mycophenolic acid on equimolar basis
  Other Names: EC-MPS

SUMMARY:
The purpose of this study is to learn more about symptoms and gastrointestinal lesions associated with taking myfortic® by switching patients to a delayed release formulation that is developed to alleviate GI symptoms. A comparison of the frequency and severity of GI symptoms observed in patients treated with MMF (cellcept®) after conversion to myfortic® will be measured by using a self-assessed questionnaire called Gastrointestinal Symptom Rating Scale (GSRS). To prove the incidence and improvement of GI lesions in patients treated with MMF (cellcept®) after conversion to myfortic® will be measured by using Small Bowel Capsule Endoscopy (SBCE).

DETAILED DESCRIPTION:
Myfortic® recently introduced to the market has shown to be similar to MMF in how effectively it works and how well it is tolerated. Both drugs have the same active ingredient, but they are different in the way that they deliver them to the body. Myfortic® is an advanced, enteric coated formulation of mycophenolate sodium (EC-MPS) that delays the release of the active ingredient, MPA. MPA has more potent effects on the lymphocytes than other cells. This makes for improved GI tolerability of the MPA therapy.

ELIGIBILITY:
Inclusion Criteria:

* Male or female patients between 18 and 75 years of age.
* Recipients of first or second cadaveric, living unrelated or living related kidney transplant.
* Recipients who are at least 4 weeks post renal transplantation with stable renal function.
* Patients who have used MMF at least 10 days and are currently receiving MMF. (up to 3g/day dosage allowed)
* Patients with at least one moderate or severe upper or lower GI complaints.
* Patients' immunosuppressive regimen other than steroids as well as medication for treatment of GI symptoms must be unchanged for at least 1 week prior to study start.
* Females of childbearing potential must have a negative pregnancy test prior to the inclusion period. Effective contraception must be used during the trial, and for 4 weeks following discontinuation of the study medication.
* Patients who are willing and able to participate in the full course of the study and from whom written informed consent has been obtained.

Exclusion Criteria:

* Multi-organ transplant patients or previous transplant with any other organ different from kidney.
* The presence of a severe GI disorder. History of a significant GI disorder prior to transplant that has remained unchanged since transplant and/or the introduction of MMF will exclude patient.
* Evidence of any GI disorder induced by an infection, underlying medical condition, or concomitant medication other than MMF.
* Modification of GI medication or MMF dose within last 1 week.
* Evidence of graft rejection, treatment of acute rejection, or unstable renal function within 4 weeks prior to the Baseline visit.
* Patients who have received an investigational immunosuppressive drug within 4 weeks prior to study entry.
* Patients with a history of malignancy within the last five years, except excised squamous or basal cell carcinoma of the skin.
* Pregnant or nursing women.
* Patients with thrombocytopenia (<75,000/mm3), with an absolute neutrophil count of <1,500/mm3 and/or leukocytopenia (<3,500/mm3), and/or hemoglobin <9.0 g/dL prior to enrollment.
* Presence of clinically significant pyrexia and/or infection requiring continued therapy.
* Evidence of severe liver disease [incl. abnormal liver profile i.e. AST, ALT or total bilirubin = 3 times the upper limit of normal].
* Patients who have any anatomical GI tract defects which have risk of capsule getting stuck such as tumor or previous abdominal surgery.
* Abnormal physical or laboratory findings of clinical significance within 2 weeks of inclusion which would interfere with the objectives of the study.
* Patients with symptoms of significant illness or evidence of current drug and/or alcohol abuse.
* Inability to self-administer the GSRS & OTE questionnaire.
* Use of other investigational drugs at the time of enrollment, or within 30 days or 5 half-lives of enrollment, whichever is longer.
* History of hypersensitivity to any of the study drugs or to drugs with similar chemical structures.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 23 (Actual)
Dates: Start 2009-04; Primary Completion 2011-03 (Actual); Study Completion 2011-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: suphamai bunnapradist, MD, Principal Investigator — University of California, Los Angeles
Locations (1):
- University of California, Los Angeles, Los Angeles, California, United States

REFERENCES:
- [Background] Shaw LM, Sollinger HW, Halloran P, Morris RE, Yatscoff RW, Ransom J, Tsina I, Keown P, Holt DW, Lieberman R, et al. Mycophenolate mofetil: a report of the consensus panel. Ther Drug Monit. 1995 Dec;17(6):690-9. doi: 10.1097/00007691-199512000-00025. No abstract available. PMID 8588243
- [Background] Ojo AO, Meier-Kriesche HU, Hanson JA, Leichtman AB, Cibrik D, Magee JC, Wolfe RA, Agodoa LY, Kaplan B. Mycophenolate mofetil reduces late renal allograft loss independent of acute rejection. Transplantation. 2000 Jun 15;69(11):2405-9. doi: 10.1097/00007890-200006150-00033. PMID 10868649
- [Background] Meier-Kriesche HU, Steffen BJ, Hochberg AM, Gordon RD, Liebman MN, Morris JA, Kaplan B. Long-term use of mycophenolate mofetil is associated with a reduction in the incidence and risk of late rejection. Am J Transplant. 2003 Jan;3(1):68-73. doi: 10.1034/j.1600-6143.2003.30112.x. PMID 12492713
- [Background] Behrend M. Adverse gastrointestinal effects of mycophenolate mofetil: aetiology, incidence and management. Drug Saf. 2001;24(9):645-63. doi: 10.2165/00002018-200124090-00002. PMID 11522119
- [Background] Salvadori M, Holzer H, de Mattos A, Sollinger H, Arns W, Oppenheimer F, Maca J, Hall M; ERL B301 Study Groups. Enteric-coated mycophenolate sodium is therapeutically equivalent to mycophenolate mofetil in de novo renal transplant patients. Am J Transplant. 2004 Feb;4(2):231-6. doi: 10.1046/j.1600-6143.2003.00337.x. PMID 14974944
- [Background] Dimenas E, Carlsson G, Glise H, Israelsson B, Wiklund I. Relevance of norm values as part of the documentation of quality of life instruments for use in upper gastrointestinal disease. Scand J Gastroenterol Suppl. 1996;221:8-13. doi: 10.3109/00365529609095544. PMID 9110389
- [Background] Kleinman L, Faull R, Walker R, Ramesh Prasad GV, Ambuehl P, Bahner U. Gastrointestinal-specific patient-reported outcome instruments differentiate between renal transplant patients with or without GI complications. Transplant Proc. 2005 Mar;37(2):846-9. doi: 10.1016/j.transproceed.2004.12.106. PMID 15848552
- [Result] Bunnapradist S, Sampaio MS, Wilkinson AH, Pham PT, Huang E, Kuo HT, Anastasi B, Danovitch GM, Lo SK. Changes in the small bowel of symptomatic kidney transplant recipients converted from mycophenolate mofetil to enteric-coated mycophenolate sodium. Am J Nephrol. 2014;40(2):184-90. doi: 10.1159/000365360. Epub 2014 Sep 2. PMID 25196230

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Kidney Transplant Clinic
Groups:
- Kidney Transplant Recipients With GI Symptoms: Small bowel capsule endoscopy (SBCE): SBCE will be performed at Day 2 and Day 30.
  Small bowel capsule endoscopy (SBCE): SBCE will be performed at Day 2.
Period: Overall Study
Arm/Group | Kidney Transplant Recipients With GI Symptoms
Started | 23
Completed | 18 (3 subjects withdrew after completing baseline questionnaire. 2 did not complete 30-day visit.)
Not Completed | 5
Not completed — Withdrawal by Subject | 3
Not completed — Lost to Follow-up | 2

BASELINE CHARACTERISTICS:
Population: of 23 participants, 18 participants completed the study.
Groups:
- Kidney Transplant Recipients With GI Symptoms: If there are negative findings on SBCE, that will be continued on MMF. No need to have second SBCE.
  Small bowel capsule endoscopy (SBCE): SBCE will be performed at Day 2 and Day 30.
  Small bowel capsule endoscopy (SBCE): SBCE will be performed at Day 2.
Arm/Group | Kidney Transplant Recipients With GI Symptoms
Number analyzed (Participants) | 18
Age, Continuous [Median (Standard Deviation); unit: years] | 45 (11.69)
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 17
  >=65 years | 1
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8
  Male | 10
Region of Enrollment [Number; unit: participants]
  United States | 18

OUTCOME MEASURES:

1. Primary Outcome: GI Mucosal Lesions Change and Clinical Symptoms Using The Gastrointestinal Symptom Rating Scale (GSRS) Score
Description: The GSRS has a seven-point graded Likert-type scale where 1 represents absence of troublesome symptoms and 7 represents very troublesome symptoms.
  A higher GSRS indicate worse symptoms and a difference between D30 and last SBCE scores greater or equal to 0.3 can be considered as a clinically significant improvement in the symptoms.
Time Frame: one month
Measure: Mean (95% Confidence Interval); unit: GSRS score
Arm/Group | Kidney Transplant Recipients With GI Symptoms
Number analyzed (Participants) | 18
GSRS score
  baseline | 2.99 [2.18 to 3.80]
  day 30 | 2.19 [1.39 to 2.99]
Statistical Analysis 1: Comparison: Kidney Transplant Recipients With GI Symptoms; The results of the initial SBCE exams were evaluated by a visually challenged GI specialist who gave us a descriptive report. By the end of the study, we submitted the final reports to the same specialist and asked his impression on the significant changes observed in patients' exams for each GI segment (stomach and small bowel). There were no comparison groups. Each patient is their own control. Given that this is a pilot study there is no power calculation; Test type: Superiority or Other; p = 0.05, t-test, 2 sided — The p value is only for GSRS score comparison only; Mean Difference (Net) = 0 — The GSRS range is 1-7

ADVERSE EVENTS:
Arm/Group | Kidney Transplant Recipients With GI Symptoms
Serious Adverse Events (participants affected / at risk) | 0/23
Other Adverse Events (participants affected / at risk) | 0/23

LIMITATIONS AND CAVEATS:
We did not enroll asymptomatic patients and in the extension of the trial the number of patients re-examined were few and the data obtained from them are not enough to provide definitive information.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No